CLINICAL TRIAL: NCT01420809
Title: Special Drug Use Investigation for ARIXTRA® (Fondaparinux) Injection
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112285
Record Dates: First submitted 2011-07-28; First posted 2011-08-22 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This post-marketing surveillance study was designed to collect and assess the information on proper use of fondaparinux injection, such as the safety and efficacy under actual use conditions, in subjects undergoing orthopedic surgery of the lower limb at high risk of developing venous thromboembolism.

(ARIXTRA® is a trademark of the GlaxoSmithKline group of companies.)

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergo orthopedic surgery of the lower limb at high risk of developing venous thromboembolism

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects undergoing orthopedic surgery of the lower limb at high risk of developing venous thromboembolism
Sampling Method: Probability Sample
Enrollment: 1280 (Actual)
Dates: Start 2007-09; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The number of incidences of adverse events in Japanese subjects undergoing orthopedic surgery of the lower limb | 3 months
Occurrence of adverse events of bleeding | 3 months
Presence or absence of venous thromboembolism after treatment of fondaparinux | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline